CLINICAL TRIAL: NCT02492685
Title: Quantificational Enhancement Pattern Analysis Using a Novel Software "Vuebox" of Contrast-enhanced Harmonic Endoscopic Ultrasonography for Differential Diagnosis Between Adenomas and Cholesterol Polyps
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study plan was cancelled because patient registration was delayed for the trials.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0033
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Gallbladder Polyp
Keywords: Quantitative analysis; contrast enhanced endoscopic ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast enhanced EUS group (Experimental): Contrast enhanced EUS with quantitative analysis
  Interventions: Device: Quantitative analysis by using the new developed software program VueBox

INTERVENTIONS:
Device: Quantitative analysis by using the new developed software program VueBox — After acquiring the EUS image by a regular procedure of EUS and contrast-enhanced with one of the fluoro-gas-containing contrast agents (SonoVue, Bracco, Germany), whole video is recorded on the embedded HDD (hard disk drive) of the US system for later analysis. The videos will be analyzed by using the VueBox software (Bracco Suisse SA, Geneva, Switzerland). After surgical treatment, we will compare the results of quantitative analysis with surgical pathology.

SUMMARY:
The investigators' study is a prospective study to evaluate the enhancement pattern of contrast-enhanced endoscopic ultrasonography and suggest the criterions for differential diagnosis between gallbladder polyps by using software program of quantitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* patient who will be received the exams to evaluate the polyps for treatment plan of surgical treatment
* have a plan to evaluate by EUS
* 19 years of age or older

Exclusion Criteria:

* difficult undergo EUS,
* allergy for contrast agent,
* renal failure,
* acute coronary syndrome
* pulmonary hypertension, 6) pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy between visual assessment and quantificational analysis based on surgical pathology | 1day

SECONDARY OUTCOMES:
Sensitivity between visual assessment and quantificational analysis based on surgical pathology | 1 day
Specificity between visual assessment and quantificational analysis based on surgical pathology | 1 day
PPV between visual assessment and quantificational analysis based on surgical pathology | 1 day
NPV between visual assessment and quantificational analysis based on surgical pathology | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei Institute of Gastroenterology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Wildner D, Pfeifer L, Goertz RS, Bernatik T, Sturm J, Neurath MF, Strobel D. Dynamic contrast-enhanced ultrasound (DCE-US) for the characterization of hepatocellular carcinoma and cholangiocellular carcinoma. Ultraschall Med. 2014 Dec;35(6):522-7. doi: 10.1055/s-0034-1385170. Epub 2014 Sep 9. PMID 25202903
- [Background] Saftoiu A, Vilmann P, Dietrich CF, Iglesias-Garcia J, Hocke M, Seicean A, Ignee A, Hassan H, Streba CT, Ioncica AM, Gheonea DI, Ciurea T. Quantitative contrast-enhanced harmonic EUS in differential diagnosis of focal pancreatic masses (with videos). Gastrointest Endosc. 2015 Jul;82(1):59-69. doi: 10.1016/j.gie.2014.11.040. Epub 2015 Mar 16. PMID 25792386